CLINICAL TRIAL: NCT00365638
Title: Effects of Simvastatin on Clinical, Endocrine, Metabolic and Biochemical Parameters of Women With Polycystic Ovary Syndrome: Prospective, Randomized Trial.
Brief Title: Simvastatin Therapy in Women With Polycystic Ovary Syndrome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Collaborators: Yale University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 636/04
Record Dates: First submitted 2006-08-15; First posted 2006-08-17 (Estimated); Last update posted 2006-08-17 (Estimated); Status verified 2004-09

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PCOS; statin; testosterone; lipids
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Simvastatin

INTERVENTIONS:
Drug: simvastatin

SUMMARY:
The purpose of this study is to determine whether statins (simvastatin) improve clinical (excessive hair, skin problems), endocrine (androgens) and metabolic (lipids, markers of systemic inflammation) in women with polycystic ovary syndrome (PCOS).

ELIGIBILITY:
Inclusion Criteria:

* PCO - ESHRE/ASRM criteria: oligomenorrhea (<8 spontaneous menses per year) and hyperandrogenism (hirsutism or acne) or hyperandrogenemia (testosterone >70ng/dl)
* Normal prolactin, TSH, 17-OH progesterone
* No evidence of androgen producing malignancy, Cushing's syndrome or acromegaly
* Age 18-40
* Reliable use of birth control pill for at least 3 months and no plans of pregnancy

Exclusion Criteria:

* Elevated creatinine kinase above 2 times upper limit of normal or liver enzymes (transaminases) above 2 times of upper limit of normal
* Use of any of the following medications: cyclosporine, fibrates, niacin, antifungal agents, macrolide antibiotics.
* Use of oral contraceptives and other steroid hormones 3 months prior to the study
* Contraindications to oral contraceptives

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2004-04; Study Completion 2005-02

PRIMARY OUTCOMES:
serum testosterone

SECONDARY OUTCOMES:
serum lutropin
serum follitropin
serum lipids
serum DHEA-S
serum SHBG
serum insulin

CONTACTS AND LOCATIONS:
Overall Officials: Leszek Pawelczyk, MD PhD, Principal Investigator — Poznan University of Medical Sciences; Antoni J Duleba, MD, Study Director — Yale University
Locations (1):
- Division of Infertility and Reproductive Endocrinology, Department of Gynecology and Obsterics, Poznan, Poland

REFERENCES:
- [Result] Duleba AJ, Banaszewska B, Spaczynski RZ, Pawelczyk L. Simvastatin improves biochemical parameters in women with polycystic ovary syndrome: results of a prospective, randomized trial. Fertil Steril. 2006 Apr;85(4):996-1001. doi: 10.1016/j.fertnstert.2005.09.030. Epub 2006 Mar 9. PMID 16580386
- [Derived] Xiong T, Fraison E, Kolibianaki E, Costello MF, Venetis C, Kostova EB. Statins for women with polycystic ovary syndrome not actively trying to conceive. Cochrane Database Syst Rev. 2023 Jul 18;7(7):CD008565. doi: 10.1002/14651858.CD008565.pub3. PMID 37462232
- [Derived] Banaszewska B, Pawelczyk L, Spaczynski RZ, Dziura J, Duleba AJ. Effects of simvastatin and oral contraceptive agent on polycystic ovary syndrome: prospective, randomized, crossover trial. J Clin Endocrinol Metab. 2007 Feb;92(2):456-61. doi: 10.1210/jc.2006-1988. Epub 2006 Nov 14. PMID 17105841